CLINICAL TRIAL: NCT07395947
Title: Adolescent Elite Athletes: A Comparative Biomechanical Study of Trunk Mobility, Lower Extremity Flexibility, and Functional Balance Across Sports Branches
Brief Title: Adolescent Elite Athletes: Trunk Mobility, Lower Extremity Flexibility, and Functional Balance Across Sports
Acronym: TEF-BALANCE
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: TU-SBF-2025-10-27
Record Dates: First submitted 2025-12-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Functional Balance; Mobility Limitation; Lower Extremity Problem
Keywords: Adolescent Athletes; balance; lower extremity
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Wrestling Athletes Group/ Cohort: Elite male adolescent athletes competing in wrestling.
  Interventions: Other: No intervention
- Sprint Athletes Group/ Cohort: Elite male adolescent athletes competing in sprint athletics.
  Interventions: Other: No intervention
- Canoe/Kayak Athletes Group/ Cohort: Elite male adolescent athletes competing in canoe/kayak disciplines.
  Interventions: Other: No intervention
- Taekwondo Athletes Group/ Cohort: Elite male adolescent athletes competing in taekwondo.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was administered. This study was observational in nature

SUMMARY:
This cross-sectional observational study compared trunk mobility, hamstring flexibility, and dynamic functional balance performance among elite male adolescent athletes aged 15-17 years from different sports branches, including wrestling, sprint athletics, canoe/kayak, and taekwondo.

All assessments were conducted during a single baseline evaluation session using standardized, non-invasive clinical measurement tools. Trunk mobility was assessed using a digital inclinometer, hamstring flexibility was evaluated with the passive Straight Leg Raise test using a goniometer, and dynamic functional balance was measured using the Y-Balance Test composite score on the dominant lower extremity.

The findings of this study provide sport-specific reference data and contribute to the identification of biomechanical characteristics related to mobility, flexibility, and balance in elite adolescent athletes across different sports disciplines.

DETAILED DESCRIPTION:
This study was conducted as a cross-sectional observational investigation in elite male adolescent athletes aged 15-17 years who were actively training and competing in different sports branches, including wrestling, sprint athletics, canoe/kayak, and taekwondo. The study aimed to compare trunk mobility, hamstring flexibility, and dynamic functional balance performance across different sports disciplines and to identify sport-specific biomechanical characteristics in this population.

All participants underwent a single baseline assessment at study enrollment. Trunk mobility was evaluated using a digital inclinometer to measure active spinal flexion, extension, and rotation at the lumbosacral and thoracolumbar regions. Hamstring flexibility was assessed on the dominant lower extremity using the passive Straight Leg Raise test with a clinical goniometer. Dynamic functional balance was assessed using the Y-Balance Test, and a normalized composite score was calculated based on anterior, posteromedial, and posterolateral reach distances.

Demographic and training-related characteristics, including age, training history, sport branch, and dominant limb, were recorded for descriptive purposes. Body composition parameters, including body fat percentage and body mass index, were obtained for participant profiling only and were not analyzed as primary study outcomes.

All assessments were non-invasive and were performed by an experienced physiotherapist using standardized clinical protocols. The findings of this study are expected to provide sport-specific reference values, support performance evaluation, and contribute to injury risk awareness and biomechanical profiling in elite adolescent athlete populations.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Male adolescent athletes aged 15-17 years
* Licensed and actively training and competing in their respective sports branch
* Minimum of 3 years of continuous training experience
* Ability to complete all clinical and biomechanical assessments
* Written informed consent obtained from the participant and a parent or legal guardian

Exclusion Criteria:

* Acute musculoskeletal injury within the past 3 months
* Chronic lower extremity or spinal pathology
* History of orthopedic surgery within the past 6 months
* Neurological, metabolic, or systemic condition affecting movement or balance
* Inability to comply with the testing protocol or incomplete assessment data

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male elite sprinter athletes
Study Population: The study population consists of elite male adolescent athletes aged 15-17 years who are actively training and competing in different sports branches, including wrestling, sprint athletics, canoe/kayak, and taekwondo. Participants are recruited from sports performance centers and evaluated using standardized, non-invasive clinical assessments of trunk mobility, flexibility, and functional balance.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Y-Balance Test Composite Score (%) | At study enrollment (single baseline assessment)
  Dynamic functional balance performance assessed using the Y-Balance Test. The composite score is calculated from normalized anterior, posteromedial, and posterolateral reach distances performed on the dominant lower extremity.

SECONDARY OUTCOMES:
Trunk Mobility - Inclinometer Range of Motion (°) | At study enrollment (single baseline assessment)
  Spinal mobility assessed using a digital inclinometer. Active trunk flexion, extension, and rotation angles are measured at the lumbosacral and thoracolumbar regions and recorded in degrees on the dominant side.
Hamstring Flexibility - Straight Leg Raise Angle (°) | At study enrollment (single baseline assessment)
  Hamstring flexibility evaluated using the passive Straight Leg Raise test on the dominant lower extremity. The maximum tolerated hip flexion angle is measured in degrees using a clinical goniometer.
Body Fat Percentage (%) | At study enrollment (single baseline assessment)
  Body fat percentage measured using a multi-frequency bioelectrical impedance analysis device. This parameter is collected for descriptive and profiling purposes only.
Body Mass Index (BMI, kg/m²) | At study enrollment (single baseline assessment)
  Body mass index calculated as body weight divided by height squared (kg/m²). BMI is collected for descriptive and participant profiling purposes only.

CONTACTS AND LOCATIONS:
Overall Officials: burcin ugur tosun, Study Chair — Ministry of Youth and Sports, Olympic Preparation Center, Adana, Türkiye
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus